CLINICAL TRIAL: NCT03638726
Title: Combined Subconjunctival Atropine and Intracameral Epinephrine Injection for Pupil Dilation in Phacoemulsification Under Peribulbar Anesthesia.
Brief Title: Subconjunctival Atropine and Intracameral Epinephrine for Pupil Dilation in Phacoemulsification
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ashraf Nossair, MD, Associate Professor of Ophthalmology, Cairo University, Dar El Oyoun Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 00001211
Record Dates: First submitted 2018-02-05; First posted 2018-08-20 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Cataract; Mydriasis; Adverse Drug Event
Keywords: intraoperative mydriasis; subconjunctival atropine; intracameral epinephrine; cataract surgery
MeSH Terms: conditions — Cataract; Mydriasis; Drug-Related Side Effects and Adverse Reactions | interventions — Atropine; Epinephrine; Cyclopentolate; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Randomized clinical study
Who Masked: Outcomes Assessor
Masking Description: Preoperative and postoperative assessment will be done by a masked observer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atropine sulfate and Epinephrine (Experimental): Perioperative pupil dilation is achieved by combined use of subconjunctival Atropine sulfate 0.6 mg ( parasympathetic antagonist) and intracameral Epinephrine 1:100000 ( sympathetic agonist).
  Interventions: Drug: Atropine sulfate and epinephrine
- Topical cyclopentolate and phenylephrine (Other): Preoperative pupil dilation was achieved using topical cyclopentolate and phenylephrine.
  Interventions: Drug: Topical cyclopentolate and phenylephrine

INTERVENTIONS:
Drug: Atropine sulfate and epinephrine — Experimental arm:Combined use of subconjunctival atropine sulfate 0.6 mg ( parasympathetic antagonist) and intracameral epinephrine 1:100000 ( sympathetic agonist). Control arm :topical mydriatics are used for pupil dilation.
  Other Names: Atropine (Misr.co), Epinephrine (Misr.co)
  Arms: Atropine sulfate and Epinephrine
Drug: Topical cyclopentolate and phenylephrine — Control arm: Preoperative cyclopentolate and phenylephrine eye drops are used.
  Other Names: Cyclophrine eye drops
  Arms: Topical cyclopentolate and phenylephrine

SUMMARY:
Mydriatic eye drops are routinely used before phacoemulsification but they are not free of drawbacks. Several alternatives were tried to overcome their limitations.

DETAILED DESCRIPTION:
The study will include 20 patients with bilateral cataract (40 eyes). The experimental group will include eyes for which a new injectable mydriatic combination are used to dilate the pupil. The control group will include cases where standard mydriatic eye drops are used.

ELIGIBILITY:
Inclusion Criteria:

* Cases of bilateral visually significant cataract

Exclusion Criteria:

* Poor pupil dilation(less than 6 mm diameter).
* History of previous eye surgery or trauma
* History of use of eye drops affecting pupil size such as pilocarpine.
* Known drug allergy to cyclopentolate,phenylephrine, atropine sulfate or epinephrine.
* Pediatric age group (less than 18 years old).
* Pupil abnormalities, such as anisocoria or neurological disorders.
* Associated glaucoma, uveitis, corneal, retinal or optic nerve disease.
* Cases scheduled for phacoemulsification under general anaesthesia (to exclude possible ocular and systemic effects or interactions of anaesthetic agents).
* Patients with bleeding tendency or on anti-coagulant therapy (because peribulbar and subconjunctival injections are used).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pupil diameter | 1 day
  Intraoperative pupil diameter measurements of involved eye in mm

SECONDARY OUTCOMES:
Postoperative complications | Starting from first postoperative day till one month.
  Complications such as subconjunctival hemorrhage or corneal edema
  [Time Frame: starting from the first postoperative day till one month]
Postoperative corneal thickness | 1 month after surgery
  Measured by specular microscopy in ( mm )
Postoperative corneal endothelial density | 1 month after surgery
  Measured by specular microscopy in ( cell number/mm2)
Postoperative pupil diameter | one day, one week and one month after surgery
  Postoperative diameter of involved eye in mm
Postoperative visual acuity | One day, one week and one month after surgery
  Postoperative best corrected distance visual acuity in logmar units.
Postoperative intraocular pressure (IOP) | One day, one week and one month after surgery
  Postoperative IOP measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Nossair, Principal Investigator — Dar El Oyoun Hospital
Locations (1):
- Dar El Oyoun Hospital, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Identity and names of participant will be hidden. Data related to outcome measures can be shared